CLINICAL TRIAL: NCT02858323
Title: Complement (C1q) Binding to HLA Antibodies in a Solid-Phase Immunoassay and Clinical Effect on Platelet Transfusion
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Other Study IDs: 999916155; 16-CC-N155
Record Dates: First submitted 2016-08-04; First posted 2016-08-08 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2025-09-10

CONDITIONS: Thrombocytopenia; Platelet Transfusion Refractoriness
Keywords: Alloimmunization; Refractoriness; Corrected Count Increment; HLA-Compatible; Natural History
MeSH Terms: conditions — Thrombocytopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Previously selected HLA-alloimmunized platelet refractory, clinical, patients.

SUMMARY:
Background:

Platelets are blood cells that help blood clot. Some people have what is called thrombocytopenia. This means they have a low blood platelet count. They need platelet transfusions very often. Human leukocyte antigen (HLA) alloimmunization occurs for a lot of these people. They become refractory. This means their platelet levels no longer increase after transfusions. Researchers want to study a procedure that detects HLA antibodies. They want to test how well it predicts how a person will respond to a transfusion. They want to see if it does this better than the procedure that is usually used.

Objective:

To study the effect of C1q-binding of Class I HLA antibodies on platelet refractoriness in people who get platelet transfusions. To test if this method better predicts response to platelet transfusion than the IgG solid phase immunoassay method.

Eligibility:

People enrolled on protocols 11-C-0136, 08-H-0156, 03-C-0277, 01-C-0157, or 01-C-0129 who:

Agreed to have their specimens and data used for future research

Had Class I HLA antibodies detected by the IgG method

Had one or more platelet transfusions at NIH after the first positive HLA IgG antibody result

Design:

For each participant, researchers will look at a small portion of their archived plasma sample. The samples were left over from prior HLA antibody tests.

Participants samples will be analyzed. They will be tested to see if C1q-binding HLA antibodies are present. This will be done by solid phase immunoassay. Results will be compared with the past results of the IgG method.

Participants data will be stored in database that s protected by password.

DETAILED DESCRIPTION:
Human leukocyte antigen (HLA) alloimmunization is common in patients undergoing frequent platelet transfusion, and is the most important cause of immune platelet refractoriness. Management strategies in HLA alloimmune platelet-refractory patients include transfusion with HLA-matched or crossmatched platelets; however, in broadly-sensitized patients, or in patients with uncommon HLA types, antigen-negative or epitope compatible donors may be difficult to find.

The Luminex immunoglobulin (Ig)G single-antigen-bead (SAB) solid phase immunoassay is now commonly used to detect HLA antibodies. However, an assay that specifically detects C1qbinding to HLA antibodies has been reported to identify a clinically relevant subset of HLA antibodies in solid organ transplantation; one group has studied the utility of this assay in platelet transfusion of HLA-alloimmunized platelet refractory patients. We intend to evaluate the ability of this C1-binding immunoassay to predict response to platelet transfusion in HLA alloimmune patients.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Class I HLA antibodies detected by the IgG solid phase immunoassay method
  2. Greater than or equal to 1 episode of platelet transfusion at NIH after the first positive HLA IgG antibody result

EXCLUSION CRITERIA:

1) Hyperproliferative thrombocytopenia

Ages: 3 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2016-07-27; Primary Completion 2017-06-20 (Actual); Study Completion 2017-06-20 (Actual)

PRIMARY OUTCOMES:
Corrected count increment after platelet transfusion | Retrospective
  Corrected Count Increment

CONTACTS AND LOCATIONS:
Overall Officials: Willy A Flegel, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Chen G, Sequeira F, Tyan DB. Novel C1q assay reveals a clinically relevant subset of human leukocyte antigen antibodies independent of immunoglobulin G strength on single antigen beads. Hum Immunol. 2011 Oct;72(10):849-58. doi: 10.1016/j.humimm.2011.07.001. Epub 2011 Jul 18. PMID 21791230
- [Background] Fontaine MJ, Kuo J, Chen G, Galel SA, Miller E, Sequeira F, Viele M, Goodnough LT, Tyan DB. Complement (C1q) fixing solid-phase screening for HLA antibodies increases the availability of compatible platelet components for refractory patients. Transfusion. 2011 Dec;51(12):2611-8. doi: 10.1111/j.1537-2995.2011.03194.x. Epub 2011 May 26. PMID 21615749
- [Background] Loupy A, Lefaucheur C, Vernerey D, Prugger C, Duong van Huyen JP, Mooney N, Suberbielle C, Fremeaux-Bacchi V, Mejean A, Desgrandchamps F, Anglicheau D, Nochy D, Charron D, Empana JP, Delahousse M, Legendre C, Glotz D, Hill GS, Zeevi A, Jouven X. Complement-binding anti-HLA antibodies and kidney-allograft survival. N Engl J Med. 2013 Sep 26;369(13):1215-26. doi: 10.1056/NEJMoa1302506. PMID 24066742